# Statistical Analysis Plan

#### **Document Control**

Title: Statistical Analysis Plan for the Study of SGLT2 Inhibitors in Lupus Nephritis Patients

Protocol ID: [NCT05748925]

Version: 1.0

Date: [11/3/2024]

Principal Investigator: [Nourelsabah Mohamed Elbialy]

Statistician: [Nourelsabah Mohamed Elbialy]

Approval Signatures:

Principal Investigator: Nourelsabah Mohamed Elbialy

Statistician: Nourelsabah Mohamed Elbialy

### **Table of Contents**

- 1. Introduction
- 2. Study Design
- 3. Study Objectives
- 4. Endpoints
- 5. Sample Size Justification
- 6. Statistical Methods
- 7. Handling of Missing Data
- 8. Interim Analysis
- 9. Safety Analysis
- 10. **Data Quality and Management**
- 11. **Software**
- 12. **Appendices**

### 1. Introduction

 Purpose of the SAP: This document outlines the statistical approach for analyzing data from the clinical trial studying the effects of SGLT2 inhibitors on renal, cardiovascular, and hematological outcomes in lupus nephritis patients.

## 2. Study Design

**Design:** Randomized, double-blind, placebo-controlled clinical trial.

Study Duration: Conducted from September 2022 to November 2023

**Randomization**: Patients were randomly assigned to either dapagliflozin (10 mg once daily) or placebo groups using computer-generated random tables in a 1:1 ratio stratified by age and gender.

**Blinding:** The study was double-blinded, and all trial staff and participants remained unaware of individual treatment assignments until study completion.

# 3. Study Objectives

**Primary Objective:** To evaluate the impact of SGLT2 inhibitors on renal, cardiovascular, and hematological parameters in lupus nephritis patients.

**Secondary Objective:** To explore changes in body weight, BMI, and other echocardiographic and iron profile parameters over 12 months.

## 4. Endpoints

**Primary Endpoints** 

Renal Function: Serum creatinine, eGFR, and 24-hour urine protein

Cardiovascular Health: BNP levels and coronary calcification via NCCT

Hematological Parameters: Hemoglobin and erythropoietin levels

Hepcidin Level: Measured before and after intervention

**Secondary Endpoints** 

Body Weight and BMI: Assessed at baseline and follow-up visits.

**Echocardiographic Findings:** Assessed pre- and post-intervention.

Iron Profile: Serum ferritin and TSAT

### 5. Sample Size Justification

**Calculation**: A sample size of 100 patients was targeted, accounting for potential dropouts, to provide sufficient power (80%) at a significance level of 0.05 to detect differences between the two groups.

### 6. Statistical Methods

#### **General Considerations**

**Significance Level:** A two-sided alpha level of 0.05 will be used for all primary analyses.

Analysis Populations:

**Intent-to-Treat (ITT):** All randomized patients will be analyzed according to their assigned group.

**Per-Protocol (PP):** Only patients completing the study without major protocol violations.

#### **Primary Endpoint Analysis**

**Renal Outcomes:** ANOVA for repeated measures for serum creatinine and eGFR if normally distributed, and the Friedman test for non-normally distributed data. Post-hoc tests using Bonferroni correction.

**Cardiovascular Outcomes:** Mann-Whitney U test for BNP levels and coronary calcification between groups.

**Hematological Outcomes:** Paired t-test for hemoglobin and erythropoietin levels if data is normally distributed; otherwise, Wilcoxon signed-rank test.

#### **Secondary Endpoint Analysis**

Body Weight and BMI: Compared over time using ANOVA for repeated measures.

**Echocardiographic Parameters:** Analyzed with paired t-tests, adjusted with Bonferroni correction.

**Iron Profile:** Analyzed pre- and post-intervention using ANOVA or Kruskal-Wallis for non-normally distributed variables.

#### **Categorical Variables**

**Chi-Square Test:** For between-group comparisons of categorical data (e.g., presence of diabetes, hypertension).

# 7. Handling of Missing Data

**Imputation:** Last observation carried forward (LOCF) for data missing at random; multiple imputation for extensive missing data.

**Sensitivity Analysis:** Conducted to evaluate the robustness of primary endpoint findings against different missing data assumptions.

## 8. Interim Analysis

**Timing:** An interim analysis is planned at the halfway point (6 months).

**Stopping Rules:** An O'Brien-Fleming approach will be applied to adjust the significance threshold for interim testing, allowing for an earlier stop for efficacy or safety concerns.

### 9. Safety Analysis

**Adverse Events (AEs):** Summarized by type, frequency, and severity. Fisher's exact test will be used to compare AE rates between groups.

**Specific Safety Parameters:** Monitoring for hypotension, electrolyte imbalances, and kidney function.

# 10. Data Quality and Management

**Data Quality Measures:** Includes data verification, regular audits, and query resolution.

Database Lock: Data will be locked and verified prior to the final analysis.

### 11. Software

Statistical Software: All analyses will be conducted using SPSS (Version 25).

# 12. Appendices

Table (1): Demographics and associated medical disorders:

| | Control group.<br>(n= 41) | Study group.<br>(n= 38) | P value |
|---|---|---|---|
| <b>Age (years)</b> Mean ± SD | 36.6 ± 9.6 | 38 ± 9.8 | 0.8 |
| Sex No. (%) - Male - Female | 7 (17.1%)<br>34 (82.9%) | 4 (10.5%)<br>34 (89.5%) | 0.5 |
| <b>Body weight (</b> Kg) mean ± SD | 78.9 ± 14 | 90 ± 15 | 0.5 |
| Body mass index<br>(Kg/m²) mean ± SD | 30.6 ± 10.5 | 33 ± 5.7 | 0.6 |
| Hypertension No. (%) | 37 (90.2%) | 38 (100%) | 0.1 |
| Diabetes No. (%) | 7 (17.1%) | 11 (28.9%) | 0.2 |

(Student T test or Mann-Whitney) for continuous data, and chi-square test for categorical data. Continuous data are expressed as mean (SD) or median (minimum – maximum). Categorical data are expressed as number (percentage), Level of significance < 0.05.

**Table (2): SLE characteristics:** 

| | Control group.<br>(n=41) | Study group.<br>(n= 38) | P value |
|---|---|---|---|
| <b>Disease duration</b> (years)<br>Median (min, max) | 6 (1, 20) | 7(1,19) | 0.3 |

| Lupus nephritis class No. (%) - Class I - Class III - Class IV - Class V - Class VI | 1 (2.4%)<br>2 (4.9%)<br>11 (26.8%)<br>26 (36.4%)<br>5 (2.4%)<br>0 (0%) | 1 (2.6%)<br>7 (18.4%)<br>8 (21.1%)<br>16 (42.1%)<br>1 (13.2%)<br>1 (2.6%) | 0.1 |
|---|---|---|---|
| Activity index Median (min, max) | 6 (0, 19) | 6 (0, 21) | 0.8 |
| Chronicity index Median (min, max) | 2 (0, 8) | 5 (0, 14) | 0.2 |
| Anti- phospholipid No. (%) | 6 (14.6%) | 3 (7.9%) | 0.4 |
| Immunosuppressive medications No. (%) - Steroid + MMF - Steroid + CNI - Steroid + CNI + MMF - Steroid + Azathioprine - Steroid | 27 (65.9%)<br>5 (12.2 %)<br>2 (4.9 %)<br>7 (17.1%)<br>0 (0%) | 18 (47.4%)<br>4 (10.5%)<br>1 (2.6%)<br>14 (36.8%)<br>1 (2.6%) | 0.2 |
| Cyclophosphamide No. (%) | 7 (17.1%) | 5 (13.2%) | 0.7 |
| Other medications No. (%) - Aspirin - Statins - Allopurinol - ACEI/ARBS - Diuretics | 15 (36.6%)<br>30 (73.2%)<br>10 (24.4%)<br>26 (63.4%)<br>14 (34.1%) | 18 (34.4%)<br>24 (63.2%)<br>14 (36.8%)<br>27(71.1%)<br>16 (32.1%) | 0.3<br>0.4<br>0.3<br>0.4<br>0.3 |

<sup>-</sup> MMF: mycophenolate mofetil; CNI: calcineurin inhibitors; ACEI/ARBS: angiotensin converting enzyme inhibitors/angiotensin receptor blockers; (Student T test or Mann-Whitney) for continuous data, and chi-square test for categorical data. Continuous data are expressed as mean (SD) or median (minimum – maximum). Categorical data are expressed as number (percentage).; Level of significance < 0.05.

**Table (3): Baseline laboratory investigations:** 

| | Control group.<br>(n= 41) | Study group.<br>(n= 38) | P value |
|---|---|---|---|
| Consumed C3 & C4<br>No. (%) | 5 (12.2%) | 2 (5.3%) | 0.4 |

| S. creatinine<br>(mg/dL) Median<br>(min, max) | 0.8 (0.4, 2.7) | 0.8 (0.4, 2.6) | 0.8 |
|---|---|---|---|
| <b>24- hour urinary protein</b> (g/24 hours) mean ± SD | 0.4 (0.06-3.6) | 0.6 (0.07-3) | 0.3 |
| eGFR (ml/min/m²)<br>mean ± SD | 114 ± 51 | 128 ± 59.7 | 0.6 |
| <b>Cholesterol</b> mg/dL mean ± SD | 185 ± 46 | 172 ± 40.7 | 0.5 |
| <b>Albumin</b> (g/dL) mean ± SD | 3.7 ± 0.4 | 3.7 ± 0.3 | 0.4 |
| Random blood<br>sugar (mg/dL)<br>Median (min, max) | 89 (66, 568) | 92.5 (64, 243) | 0.4 |
| Uric acid (mg/dL)<br>mean ± SD | 6.2 ± 2.1 | 6.5 ± 1.7 | 0.2 |
| Alanine<br>aminotransferase<br>(IU/L) Median (min,<br>max) | 17 (2, 84) | 17 (7, 82) | 0.8 |
| Aspartate<br>aminotransferase<br>(IU/L) Median (min,<br>max) | 21(9, 66) | 19 (12,72) | 0.4 |
| <b>Sodium</b> (mEq/L) mean ± SD | 137 ± 3.1 | 136 ± 3 | 0.5 |
| Potassium (mEq/L) mean ± SD | 3.9 ± 0.4 | 4 ± 0.4 | 0.3 |

eGFR: estimated glomerular filtration rate; (Student T test or Mann-Whitney) for continuous data, and chi-square test for categorical data. Continuous data are expressed as mean (SD) or median (minimum – maximum). Categorical data are expressed as number (percentage). Level of significance < 0.05.

Table (4): Baseline hematological findings:

| | Control group.<br>(n=41) | Study group.<br>(n= 38) | P value |
|---|---|---|---|
| <b>Hemoglobin</b> (g/dL)<br>Mean ± SD | $11.9 \pm 1.9$ | $11.7 \pm 1.7$ | 0.5 |
| MCV (FL) Mean ± SD | 82 ± 7 | $84 \pm 6.9$ | 0.9 |
| MCH (Pg) Mean ± SD | $25.4 \pm 2.9$ | $26.3 \pm 2.9$ | 0.9 |
| Ferritin (mg/dL)<br>Median (min, max) | 60 (13, 1113) | 33.5 (3, 1460) | 0.09 |
| TSAT (%) Median (min, max) | 23.8 (7, 64) | 18 (6, 74) | 0.05 |
| Erythropoietin<br>level (IU/L) Mean ±<br>SD | $11.6 \pm 2.1$ | $11.3 \pm 1.4$ | 0.1 |
| Hepcidin level (ug/L) Mean ± SD | 198 ± 74 | 182 ± 76 | 0.3 |
| Platelet count (*10 <sup>3</sup> )<br>Mean ± SD | 288 ± 71 | $300 \pm 79$ | 0.7 |

MCV: Mean corpuscle volume; MCH: Mean corpuscular hemoglobin; TSAT: Transferrin saturation test; (Student T test or Mann-Whitney) for continuous data, and chi-square test for categorical data. Continuous data are expressed as mean (SD) or median (minimum – maximum). Categorical data are expressed as number (percentage).; Level of significance < 0.05.

**Table (5): Baseline Cardiac evaluation:** 

| C41 | C4 | D I |
|----------------|--------------|---------|
| Control group. | Study group. | P value |

| | (n=41) | (n=38) | |
|---|---|---|---|
| Coronary calcification No. | 3 (7.3%) | 11 (28.9%) | 0.012 |
| Coronary calcification severity No. (%) - No - Minimal - Mild - moderate | 38 (92.7%)<br>1 (2.4%)<br>1 (2.4%)<br>1 (2.4%) | 27 (71.1%)<br>3 (7.9%)<br>7 (18.4%)<br>1 (2.6%) | 0.04 |
| BNP (ng/L)<br>Median (min,<br>max) | 52 (40, 557) | 52 (34, 90) | 0.8 |
| Echocardiographic | | | |
| EF % Mean ± SD | $65.4 \pm 9.3$ | $64.6 \pm 5.4$ | 0.6 |
| LAD (ml) Mean ± SD | $24.2 \pm 7.6$ | $24.9 \pm 7.6$ | 0.6 |
| Aortic diameter (ml) Mean ± SD | 24.7±7.4 | 24.8±7.1 | 0.9 |
| ESV (ml/m)<br>Median (min,<br>max) | 38±13.6 | 41±13.9 | 0.4 |
| $\begin{array}{c} \textbf{EDV} & (ml/m) \\ Mean \pm SD \end{array}$ | 98±35.7 | 111.5±31.6 | 0.08 |

BNP: Brain natriuretic peptide; EF: Ejection fraction; LAD: Left atrial dimension; ESV: End-systolic volume; EDV: End diastolic volume; (Student T test or Mann-Whitney) for continuous data, and chi-square test for categorical data. Continuous data are expressed as mean (SD) or median (minimum – maximum). Categorical data are expressed as number (percentage).; Level of significance < 0.05.

**Table (6)**: Comparison between study and control groups as regard effect of intervention on disease activity and renal affection at different time points

| | Grouping | Baseline | 3<br>months | 6 months | 9 months | 12 months | P value* |
|---|---|---|---|---|---|---|---|
| Consumed C3 & C4 | Control | 5 (12.2%) | 5<br>(12.2%) | 4 (9.8%) | 6 (14.6%) | 10 (24.4%) | 0.1 |
| No. (%) | Study | 2 (5.3%) | 5<br>(13.2%) | 2 (5.3%) | 6 (15.8%) | 6 (15.8%) | 0.1 |
| | P value** | 0.4 | 0.9 | 0.3 | 1 | 0.4 | |
| S. creatinine (mg/dL) | Control | 0.8 (0.4,<br>2.7) | 0.9 (0.4,<br>3.1) | 0.9 (0.3-<br>3.1) | 0.9 (0.6, 4) | 0.9 (0.6, 5) | 0.1 |
| Median (min, max) | Study | 0.8 (0.4,<br>2.6) | 0.9 (0.6,<br>2.6) | 0.9 (0.5,<br>3.1) | 1 (0.5,<br>4.2)<br>a | 0.9 (0.5, 5) | 0.01 |
| | P value** | 0.8 | 0.8 | 1 | 0.5 | 0.8 | |
| eGFR (ml/min/m²) | Control | 114±51 | 104±45<br>a | 107±53.8 | 99±47<br>a | 100.3±44.5<br>a | 0.003 |
| Mean ± SD | Study | 128±59.7 | 115±47<br>A | 118±50<br>A | 109±44.5<br>a, c | 115.7±48<br>a | 0.001 |
| | P value** | 0.6 | 0.9 | 0.8 | 0.2 | 0.9 | |
| | Control | 0.4(0.06-<br>3.6) | 0.6<br>(0.03-5) | 0.6 (0.03-<br>7) | 0.6 (0.02,<br>5) | 0.5 (0.02,<br>8) | 0.06 |
| <b>24- hour urinary protein</b> (g/24 hours) Median (min, max) | Study | 0.6<br>(0.07-3) | 0.7<br>(0.01-4) | 0.8 (0.02,<br>4.8) | 0.6 (0.05,<br>4.7) | 0.5 (0.02,<br>4) | 0.07 |
| | P value** | 0.3 | 0.9 | 0.8 | 0.6 | 0.6 | |
| Albumin (g/dL) | Control | 3.7±0.4 | 3.7±0.4 | 3.6±0.4 | 3.8±0.4<br>c | 3.9±0.3<br>a, b, c | 0.001 |
| Mean ± SD. | Study | 3.7±0.3 | 3.7±0.5 | 3.7±0.3 | 3.8±0.3<br>c | 3.9±0.8<br>a, c | 0.04 |
| | P value** | 0.4 | 0.9 | 0.1 | 0.7 | 0.8 | |

<sup>(\*)</sup> Within group analysis (repeated measure ANOVA).

<sup>(\*\*)</sup> Between group analysis (Student T test or Mann-Whitney) for continuous data, and chi-square test for categorical data. Post-hoc analysis;

<sup>(</sup>a) significance against baseline <0.05; (b) significance against 3 months level <0.05, (c) significance against 6 months level <0.05, (d)

significance against 9 months level <0.05. Continuous data are expressed as mean (SD) or median (minimum – maximum). Categorical data are expressed as number (percentage).

Table (7): effect of intervention on hematological findings between both groups at different time points:

| | Grouping | Baseline | 3 months | 6 months | 9 months | 12 months | P value* |
|---|---|---|---|---|---|---|---|
| Haemoglobin<br>(g/dL) Mean ±<br>SD | Control | 11.9±1.9 | 12.2±1.9 | 11.8±2.5 | 12±1.9 | 12.2±1.9 | 0.08 |
| | Study | 11.8±1.8 | 12.3±1.7 | 12±2.5 | 11.9±2.2 | 12±2 | 0.06 |
| | P value** | 0.5 | 0.7 | 0.7 | 0.3 | 0.6 | |
| MCV (FL)<br>Mean ± SD | Control | 82±7 | 83±7 | 84±7 | 84.6±7.9 | 81.5±13 | 0.1 |
| | Study | 84±6.9 | 80±14 | 83±10 | 83.2±10.8 | 84±7 | 0.3 |
| | P value** | 0.9 | 0.1 | 0.5 | 0.5 | 0.4 | |
| MCH (Pg)<br>Mean ± SD | Control | 25.4±2.9 | 27.3±9.8 | 28.5±9 | 26.9±3.2 | 26.9±3.1 | 0.08 |
| | Study | 26.3±2.9 | 27.3±9.5 | 27±3 | 26.6±3.5 | 27.1±3.4 | 0.8 |
| (*) \( \text{\text{V}} \) | P value** | 0.9 | 0.9 | 0.4 | 0.4 | 0.5 | |

<sup>(\*)</sup> Within group analysis (repeated measure ANOVA).

MCV: Mean corpuscle volume; MCH: Mean corpuscular haemoglobin.

<sup>(\*\*)</sup> Between group analysis (Student T test or Mann-Whitney) for continuous data, and chi-square test for categorical data. Continuous data are expressed as mean (SD) or median (minimum – maximum). Categorical data are expressed as number (percentage).

| | Grouping | Baseline | 12 months | P value* |
|---|---|---|---|---|
| Ferritin (mg/dL) | Control | 60 (13, 1113) | 75 (6, 2127) | 0.5 |
| Median (min, max) | Study | 33.5 (3, 1460) | 64 (3, 1311) | 0.8 |
| | P value** | 0.09 | 0.4 | |
| TSAT (%) Median | Control | 23.8 (7, 64) | 28 (5, 62) | 0.1 |
| (min, max) | Study | 18 (6, 74) | 20 (6, 66) | 0.9 |
| | P value** | 0.05 | 0.1 | |
| Erythropoietin | Control | 11.6±2.1 | 12.8 ± 3.5 | 0.08 |
| level IU/L Mean ± SD | Study | 11.3±1.4 | 12.4 ± 3.5 | 0.1 |
| | P value** | 0.1 | 0.6 | |
| Hepcidin level ug/L | Control | 198 ± 74 | 128 ±63 | 0.001 |
| Mean ± SD | Study | 182±76 | 116±15 | 0.001 |
| | P value** | 0.3 | 0.2 | |
| Platelet count | Control | 288 ± 71 | 283 ± 74 | 0.6 |
| ( <b>×10</b> <sup>3</sup> ) Mean ± SD | Study | 300 ± 79 | 276 ± 65 | 0.01 |
| | P value** | 0.7 | 0.5 | |

<sup>(\*)</sup> Within group analysis (paired t test).

Continuous data are expressed as mean (SD) or median (minimum – maximum). Categorical data are expressed as number (percentage).

TSAT: Transferrin saturation test

Table (9): Cardiac evaluation differences between both groups after 12 months:

<sup>(\*\*)</sup> Between group analysis (Student T test or Mann-Whitney) for continuous data, and chi-square test for categorical data.

| | Control group | Study group | P value |
|---|---|---|---|
| Coronary calcification No. (%) | 1 (2.4%) | 11 (28.9%) | 0.001 |
| Coronary calcification<br>severity No. (%) - No - Minimal - Mild - moderate | 40 (97.6%)<br>0<br>0<br>1 (2.4%) | 27 (71.1%)<br>9 (23.7%)<br>2 (5.3%)<br>0 | 0.002 |
| <b>BNP</b> ng/L Mean $\pm$ Sd | $66 \pm 22.1$ | 65.8±21 | 0.9 |
| Echocardiographic findir | ıg | | |
| EF % Mean ± SD | 65.5±5.8 | 64.9±5.2 | 0.8 |
| <b>LAD</b> ml Mean $\pm$ SD | 26.7±7.6 | 28.2±8.6 | 0.4 |
| <b>Aortic diameter</b> ml<br>Mean ± SD | 26.6±6.5 | 25.5±6.2 | 0.4 |
| ESV ml/min<br>Mean ± SD | 39.5±18 | 36.3±9.3 | 0.3 |
| EDV ml/min<br>Mean ± SD | 108±29.6 | 109±19.3 | 0.9 |

BNP: Brain natriuretic peptide; EF: Ejection fraction; LAD: Left atrial dimension; ESV: End- systolic volume; EDV: End diastolic volume; Chi square test; Student t- test; Man, Whitney test; Level of significance < 0.05.

Table (10): Comparison between both groups as regard post intervention side effects

| | Control group. (n=41) | Study group. (n= 38) | P value |
|---|---|---|---|
| AKI episodes No. | | | |
| - No | 38 (92.7%) | 31 (81.6%)<br>5 (13.2%) | 0.17 |
| - once | 1 (2.4%) 2 (4.9%) | 2 (5.3%) | |
| - twice | , | | |
| UTI No. (%) | | | |
| - No | 35 (85.4%)<br>4 (9.8%) | 31 (81.6%)<br>5 (13.2%) | 0.8 |
| - once | 2 (4.9%) | 2 (5.3%) | |
| - more than once | | | |
| Gynecological infection No. (%) | 1 (2.4%) | 2 (5.3%) | 0.6 |
| Viral infection No. (%) | 1(2.4%) | 1 (2.6%) | 1 |
| MMF intolerance<br>No. (%) | 1 (2.5%) | 2 (5.3%) | 0.6 |
| Renal biopsy No. (%) | 2 (4.9%) | 1 (2.6%) | 0.6 |
| Increase steroid dose No. (%) | 7 (17.1%) | 4 (10.5%) | 1 |

UTI: urinary tract infection episodes; AKI: acute kidney injury; chi-square test for categorical data. Categorical data are expressed as number (percentage).; Level of significance < 0.05.



figure1: flow chart of participating populations



Figure (2) shows difference between individual which had improved eGFR or not as regard to their basal eGFR in total cohort, which found that improving eGFR had been occurred in patients with lower eGFR ( $107\pm50 \text{ vs } 137\pm58 \text{ ml/min/m}^2$ 



**Figure (3)** show no significant difference between the drug and placebo groups (p=0.857). as regard incidence of anemia before intervention, the drug group has 23 anemic participants (60.5%) versus 24 participants (58.5%) in the placebo group, while post intervention, In the anemia category, the drug group has 16 participants (42.1%), while the placebo group has 22 participants (53.7%) with non-significant differences (p = 0.3)

Figure (4) differences in body weight between both groups at different time points:



# Glossary of Terms and Abbreviations

| AA | Amino Acids |
|------------|---------------------------------------------|
| ABIN | A20 Binding Inhibitor Of NF-Kb |
| ACE | Angiotensin-Converting Enzyme Inhibitors |
| ACR | American College of Rheumatology |
| AKI | Acute Kidney Injury |
| ALCAM | Activated Leucocyte Adhesion Molecule |
| ALP | Alkaline Phosphatase |
| AMP | Adenosine Monophosphate |
| AMPK | Amp-Activated Protein Kinase |
| ANA | Antinuclear Antibodies |
| ANG II | Angiotensin 2 |
| ANOVA | Analysis Of Variance |
| ANTI-DSDNA | Anti Double Stranded Deoxyribonucleic Acid |
| | Antibodies |
| ANTI-SM | Anti-Smith Antibodies |
| APLS | Antiphospholipid Syndrome |
| ARBS | Angiotensin 2 Receptor Blockers |
| ATN | Acute Tubular Necrosis |
| ATP | Adenosine Triphosphate |
| BAFF | B-Cell-Activating Factor |
| BLISS | B Lymphocyte Stimulator Inhibitor Belimumab |
| | Plus Standard Therapy |
| BMI | Body Mass Index |
| BNP | Brain Natriuretic Peptide |
| BP | Blood Pressure |
| CAC | Coronary Artery Calcification |
| CAD | Coronary Artery Disease |

| CAMK | Ca2+/Calmodulin-Dependent Protein Kinase |
|-----------------|------------------------------------------------|
| CASR | Serine/Threonine Kinase Camk4 |
| CCS | Coronary Calcium Score |
| CD163 | Macrophage-Specific Protein |
| CD4 T-CELLS | Helper T-Cells |
| CD8 T-CELLS | Cytotoxic T-Cells |
| CI | Confidence Interval |
| CKD | Chronic Kidney Disease |
| CKD-MBD | Chronic Kidney Disease-Mineral Bone Disorders |
| CLD | Chronic Liver Disease |
| CMV | Cytomegalovirus |
| CNI | Calcineurin Inhibitors |
| CT | Computed Tomography |
| CVD | Cardiovascular Disease |
| CYC | Cyclophosphamide |
| DAPA-HF | The Dapagliflozin and Prevention of Adverse |
| | Outcomes in Heart Failure |
| DCGF | Death-Censored Graft Failure |
| DECLARE-TIMI 58 | Dapagliflozin Effect on Cardiovascular Events- |
| | Thrombolysis in Myocardial Infarction 58 |
| DELIGHT | Delay Of Impaired Glucose Tolerance by A |
| | Healthy Lifestyle Trial |
| DM | Diabetes Mellitus |
| DNA | Deoxyribonucleic Acid |
| EBV | Epstein Bar Virus |
| EDV | End Diastolic Volume |
| EF | Ejection Fraction |
| EGFR | Estimated Glomerular Filtration Rate |
| EMPA-REG | Empagliflozin-Removing Excess Glucose |

| EPO | Erythropoietin |
|---------|-------------------------------------------|
| EPOR | Erythropoietin Receptors |
| ESRD | End-Stage Renal Disease |
| ESV | End- Systolic Volume |
| EULAR | The European League Against Rheumatism |
| FDA | Food And Drug Administration |
| FEUA | Fractional Excretion of Uric Acid |
| FGF | Fibroblast Growth Factor |
| FN1 | Fibronectin 1 |
| GCS | Glucocorticoids |
| H2 O2 | Hydrogen Peroxide |
| HBA1C | Glycated Hemoglobin |
| HBV | Hepatitis B Virus |
| HCV | Hepatitis C Virus |
| HD | Hemodialysis |
| HIF | Hypoxia-Inducible Factor |
| HIV | Human Immunodeficiency Virus |
| HLA | Human Leucocytic Antigen |
| HPT | Hyperparathyroidism |
| HR | Hazard Ratio |
| HR-PQCT | High-Resolution Peripheral Quantitative |
| | Computer Tomography |
| HUS | Hemolytic Uremic Syndrome |
| HZ | Herpes Zoster |
| IFTA | Interstitial Fibrosis and Tubular Atrophy |
| IGG | Immunoglobulin G |
| IL-6 | Interleukin-6 |
| IPTH | Intact Parathyroid Hormone |
| ITP | Immune Thrombocytopenic Purpura |

| KDIGO | Kidney Disease Improving Global Outcomes |
|--------|---------------------------------------------|
| LAD | Left Atrial Dimension |
| LDL | Low-Density Lipoprotein |
| LUMINA | Lupus In Minorities; Nature Vs. Nurture |
| LV | Left Ventricle |
| MCH | Mean Corpuscular Hemoglobin |
| MCP1 | Monocyte Chemoattractant Protein-1 |
| MCV | Mean Corpuscular Volume |
| MDCT | Multidetector CT |
| MMF | Mycophenolate Mofetil |
| MPAA | Mycophenolic Acid Analogue |
| MRI | Magnetic Resonance Imaging |
| NGAL | Neutrophil Gelatinase-Associated Lipocalin |
| NH3 | Na+/H+ Exchanger 3 |
| NHS | National Health Service |
| NLR | Nucleotide-Binding Oligomerization Domain- |
| | Like Receptor |
| NSAIDS | Non-Steroidal Anti-Inflammatory Drugs |
| PD | Peritoneal Dialysis |
| PET | Positron Emission Tomography |
| PGC-1A | Peroxisome Proliferators-Activated Receptor |
| | Gamma Coactivator-1α |
| QCT | Quantitative Computer Tomography |
| RAAS | Renin-Angiotensin-Aldosterone |
| RBG | Random Blood Glucose |
| RCTS | Randomized Controlled Trials |
| RNA | Ribonucleoside Antibodies |
| ROS | Reactive Oxygen Species |

| RPS/ISN | The Renal Pathology Society/International |
|------------------|------------------------------------------------|
| | Society of Nephrology |
| RRT | Renal Replacement Therapy |
| SBP | Systolic Blood Pressure |
| SELENA-SLEDAI | Safety Of Estrogens in Lupus Erythematosus |
| | National Assessment–SLE Disease Activity |
| | Index |
| SGLT2 | Sodium-Glucose Cotransporter 2 |
| SGLT2 inhibitors | Sodium-Glucose Cotransporter 2 Inhibitors |
| SIRT1 | Sirtuin Type 1. |
| SLE | Systemic Lupus Erythematosus |
| SLEDAI | Systemic Lupus Erythematosus Disease Activity |
| | Index |
| SLICC | The Systemic Lupus International Collaborating |
| | Clinics |
| SNS | Sympathetic Nervous System |
| T2DM | Type 2 Diabetes Mellitus |
| TLRS | Toll-Like Receptors |
| TNF | Tumor Necrosis Factor |
| TSAT | Transferrin Saturation |
| UTI | Urinary Tract Infection |
| VCAM-1 | Vascular Cell Adhesion Molecule-1 |